CLINICAL TRIAL: NCT06721208
Title: Development of a Mobile APP to Promote Physical Activity in Individuals with Knee Osteoarthritis: a "Move for Knee" Study Protocol
Brief Title: Mobile App Use for Physical Activity in Knee Osteoarthritis
Acronym: moveforknee
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Sara Liguori, doctor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0008758/i-21/03/2024
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthristis
Keywords: knee osteoarthiritis; physical activity; functioning; pain; digital health; mobile application
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): - patients who will use the "Move for Knee" APP (intervention arm);
  Interventions: Behavioral: use the "Move for Knee" APP
- control (No Intervention): patients who will be advised to engage in free physical activity (control arm).

INTERVENTIONS:
Behavioral: use the "Move for Knee" APP — The mobile APP called Move Your Knee allows the collection of data entered by patients, useful for understanding their lifestyle habits and daily physical activity level, and information relating to KOA pathology.
  At the end of the questionnaire, the algorithm integrated into the APP's computer code will allow the calculation of the patient's presumed level of physical activity. This will then be followed by the assignment of a specific form which includes the exercises and the related execution parameters (i.e. weekly frequency), and useful advice for safely carrying out the exercises to achieve the specific functional objectives.
  Arms: intervention

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of an app developed to provide useful guidance on physical activity for people with knee osteoarthritis.The main question it aims to answer is:

"What physical activity can I perform with knee osteoarthritis?" Researchers will compare use of app developed to provide physicial activity program versus educational advices (a look-alike substance that contains no drug) to see if APP works to treat pain and stiffness related to knee osteoarthritis.

Participants will:

Download and use APP Visit the clinic once every 4 weeks for checkups and tests

DETAILED DESCRIPTION:
In this no-profit, interventional, double-arm, monocentric study, men and women with unilateral or bilateral tibiofemoral KOA according to the American College of Rheumatology criteria for KOA, aged 45 to 70 years, and radiographic findings (Kellgren-Lawrence grade 1-3) referring to the Physical Medicine and Rehabilitation Unit, University of Campania "Luigi Vanvitelli", will be included. In this trial, the patients will be randomized into two groups:

* patients who will use the "Move for Knee" APP (intervention arm);
* patients who will be advised to engage in free physical activity (control arm). Patients will be directed to one of the arms through random sampling with consecutive 1:1 randomization (intervention:control).

The mobile APP called Move Your Knee is divided in 4 sections:

1. Know Your Knee: this first section allows the collection of data entered by patients, useful for understanding their lifestyle habits and daily physical activity level, and information relating to KOA pathology.

   At the end of the questionnaire, the algorithm integrated into the APP's computer code will allow the calculation of the patient's presumed level of physical activity. This will then be followed by the assignment of a specific form which includes the exercises and the related execution parameters (i.e. weekly frequency), and useful advice for safely carrying out the exercises to achieve the specific functional objectives.
2. Move Your Knee: in this section, the patient will be able to select the level of difficulty/intensity in performing the physical exercise (the more advanced levels are blocked until the previous objective is achieved).

   There are 5 levels, each marked by an evocative image that summarizes the functional meaning and, therefore, facilitates the identification of the type of user (in particular, from the most advanced level: "Hawk"; "Tiger"; "Bull", "Turtle", "Sloth").

   Once the exercise program has been started, the patient finds the indications/advice for carrying out each exercise (duration, series and repetitions). Through the motion capture function, he can record the exercise he performed, to check with your doctor the appropriateness and safety of its execution. The video obtained from this recording is saved in the APP's Database (DB) and can be transferred to the doctor via Chat.
3. Step by step: through this section, patients have the opportunity to record and monitor daily progress, obtaining a real-time view of their progress.
4. Chat: to facilitate direct contact with the doctor, the APP is equipped with a native instant messaging service, through which patients can directly contact their doctor by communicating and sharing files and videos useful for monitoring.

The system is completed with a control panel that is used by the doctor via terminal/PC. This tool allows:

1. registration of the patient on a specific web platform;
2. access to the patient files associated with the referring doctor;
3. patient monitoring, viewing the patient's progress to monitor adherence to use;
4. access to Chat. Patients will be visited at baseline corresponding to enrollment in the study (T0), and at 30 (T1), 90 (T2), and 180 days (T3).

At all time points patients will be evaluated with the following protocol:

* multidimensional pain evaluation with

  * the Brief Pain Inventory (BPI) and its two indexes (severity and interference indexes; BPI-SI, BPI-II);
  * the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale, for the neuropathic component of pain;
* stiffness and function through Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC);
* quality of life through EUROQoL-5Dimension (EQ-5D). For patients in the intervention group, questions related to the "user experience" and any adverse effects related to the APP will be included through an open-ended question "describe your experience with the APP" at 30 (T1), 90 (T2), and 180 days (T3).

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral tibiofemoral osteoarthritis according to the American College of Rheumatology classification criteria for osteoarthritis, aged between 45 and 70 years, with radiographic findings (Kellgren-Lawrence grade 1-3)
* Expression of consent to participate in the study through a signed informed consent form
* Ability to understand and use the APP through a practical demonstration in an outpatient setting

Exclusion Criteria:

* Psychiatric disorders that could potentially invalidate informed consent
* Pregnancy or breastfeeding

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) and its two indexes (severity and interference indexes; BPI-SI, BPI-II) | at 30 (T1), 90 (T2), and 180 days (T3)
  multidimensional pain evaluation

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC); | 30 (T1), 90 (T2), and 180 days (T3)
  stiffness and function
EUROQoL-5Dimension (EQ-5D). | at 30 (T1), 90 (T2), and 180 days (T3)
  quality of life

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li E, Tan J, Xu K, Pan Y, Xu P. Global burden and socioeconomic impact of knee osteoarthritis: a comprehensive analysis. Front Med (Lausanne). 2024 May 16;11:1323091. doi: 10.3389/fmed.2024.1323091. eCollection 2024. PMID 38818397
- [Background] Iolascon G, Migliore A, Beretta G, Bernetti A, Bortolotti R, Celano A, Giarratano A, Marinangeli F, Momoli A, Sebastiani GD, Tomasini A, Tonolo S, Madotto F, Di Martino A, Natoli S. Pain Management in Knee Osteoarthritis: Insights from an Exploratory Online Survey of Italian Patients and Physicians. Healthcare (Basel). 2024 Oct 18;12(20):2077. doi: 10.3390/healthcare12202077. PMID 39451492
- [Background] Geng R, Li J, Yu C, Zhang C, Chen F, Chen J, Ni H, Wang J, Kang K, Wei Z, Xu Y, Jin T. Knee osteoarthritis: Current status and research progress in treatment (Review). Exp Ther Med. 2023 Aug 25;26(4):481. doi: 10.3892/etm.2023.12180. eCollection 2023 Oct. PMID 37745043
- [Background] Lee J, Chang RW, Ehrlich-Jones L, Kwoh CK, Nevitt M, Semanik PA, Sharma L, Sohn MW, Song J, Dunlop DD. Sedentary behavior and physical function: objective evidence from the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2015 Mar;67(3):366-73. doi: 10.1002/acr.22432. PMID 25155652
- [Background] Zmerly H, Milanese C, El Ghoch M, Itani L, Tannir H, Kreidieh D, Yumuk V, Pellegrini M. Personalized Physical Activity Programs for the Management of Knee Osteoarthritis in Individuals with Obesity: A Patient-Centered Approach. Diseases. 2023 Dec 14;11(4):182. doi: 10.3390/diseases11040182. PMID 38131988
- [Background] Scopaz KA, Piva SR, Wisniewski S, Fitzgerald GK. Relationships of fear, anxiety, and depression with physical function in patients with knee osteoarthritis. Arch Phys Med Rehabil. 2009 Nov;90(11):1866-73. doi: 10.1016/j.apmr.2009.06.012. PMID 19887210